CLINICAL TRIAL: NCT01416181
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy of Natalizumab on Reducing Disability Progression in Subjects With Secondary Progressive Multiple Sclerosis, With Optional Open-Label Extension
Brief Title: A Clinical Study of the Efficacy of Natalizumab on Reducing Disability Progression in Participants With Secondary Progressive Multiple Sclerosis
Acronym: ASCEND in SPMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The ASCEND Study did not achieve statistical significance on the primary or secondary endpoints.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101MS326; 2010-021978-11 (EudraCT Number)
Record Dates: First submitted 2011-07-21; First posted 2011-08-12 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Natalizumab; secondary; multiple sclerosis; MS; SPMS; Tysabri
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Neoplasm Metastasis; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- natalizumab (Experimental): In Part 1 participants were randomized to receive 300 mg of natalizumab intravenously (IV) every 4 weeks for 96 weeks. In Part 2 participants transitioned to receive open-label natalizumab 300 mg IV every 4 weeks for at least 96 weeks.
  Interventions: Drug: natalizumab
- Placebo (Experimental): In Part 1 participants were randomized to receive placebo IV every 4 weeks for 96 weeks. In Part 2 participants transitioned to receive open-label natalizumab 300 mg IV every 4 weeks for at least 96 weeks.
  Interventions: Drug: natalizumab; Drug: Placebo

INTERVENTIONS:
Drug: natalizumab — Administered as specified in the treatment arm
  Other Names: Tysabri; BG00002
Drug: Placebo — Matched placebo in part 1
  Arms: Placebo

SUMMARY:
This is a Phase 3b, multicenter, international study conducted in 2 parts. Upon completion of the placebo-controlled period (Part 1), participants will have the option of enrolling in a 2-year open-label extension (Part 2).

Part 1: The primary objective of the study is to investigate whether treatment with natalizumab slows the accumulation of disability not related to relapses in participants with secondary progressive multiple sclerosis (SPMS).

The secondary objectives of Part 1 of this study are to determine the proportion of participants with consistent improvement in Timed 25-Foot Walk (T25FW), the change in participant-reported ambulatory status as measured by the 12-item MS Walking Scale (MSWS-12), the change in manual ability based on the ABILHAND Questionnaire, the impact of natalizumab on participant-reported quality of life using the Multiple Sclerosis Impact Scale-29 Physical (MSIS-29 Physical), the change in whole brain volume between the end of study and Week 24 using magnetic resonance imaging (MRI) and the proportion of participants experiencing progression of disability as measured by individual physical Expanded Disability Status Scale (EDSS) system scores.

Part 2: The primary objective of Part 2 of the study is to evaluate the safety profile of natalizumab in participants with SPMS.

The secondary objectives of Part 2 of the study are to investigate long-term disability (based on clinical or participant-reported assessments) in participants with SPMS receiving natalizumab treatment for approximately 4 years and to assess change in brain volume and T2 lesion volume.

ELIGIBILITY:
Key Inclusion Criteria (Part 1):

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local subject privacy regulations.
* SPMS defined as relapsing-remitting disease followed by progression of disability independent of or not explained by multiple sclerosis (MS) relapses for at least 2 years.
* EDSS score of 3.0 to 6.5, inclusive.
* Multiple Sclerosis Severity Score of 4 or higher.
* Documented confirmed evidence of disease progression independent of clinical relapses over the 1 year prior to enrollment as defined in the Study Reference Guide.

Key Exclusion Criteria (Part 1):

* Relapsing remitting multiple sclerosis (RRMS) or primary progressive MS as defined by the revised McDonald Committee criteria.
* Clinical relapse (within 3 months) prior to randomization.
* T25FW test of >30 seconds during the screening period.
* Any value below the lower limit of normal for blood levels of leukocytes, lymphocytes, or neutrophils.
* Considered by the Investigator to be immunocompromised based on medical history, physical examination, laboratory testing, or any other testing required by local guidelines, or due to prior immunosuppressive or immunomodulating treatment.
* Subjects for whom MRI is contraindicated (i.e., have pacemakers or other contraindicated implanted metal devices, are allergic to gadolinium, or have claustrophobia that cannot be medically managed).
* History of any clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (other than MS), dermatologic, psychiatric, and renal, or other major disease that would preclude participation in a clinical study.
* History of malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* Known history of or positive test result for human immunodeficiency virus.
* Positive test result for hepatitis C virus (test for hepatitis C virus antibody or hepatitis B virus (test for hepatitis B surface antigen and/or hepatitis B core antibody).
* History of transplantation or any anti-rejection therapy.
* Presence of any infectious disease (e.g., cellulitis, abscess, pneumonia, septicemia) within 30 days prior to screening.
* History of progressive multifocal leukoencephalopathy or other opportunistic infections.

Treatment History (Part 1)

* Any prior treatment with cell-depleting therapies, including total lymphoid irradiation, cladribine, rituximab, alemtuzumab, or bone marrow ablation.
* Any prior treatment with natalizumab.
* Treatment with mitoxantrone, cyclophosphamide, cyclosporine, azathioprine, methotrexate, mycophenolate mofetil, T cell or T cell receptor vaccination, fingolimod, daclizumab, or cytapheresis within 6 months prior to randomization.
* Treatment with intravenous or oral corticosteroids, intravenous immunoglobulin, or plasmapheresis for treatment of MS within the 3 months prior to randomization.
* Treatment with glatiramer acetate or any interferon beta preparations within 4 weeks prior to randomization.
* Treatment with 4-aminopyridine within 30 days prior to randomization, unless a stable dose has been maintained for at least 30 days prior to randomization and will be continued for the course of this study.

Key Inclusion Criteria (Part 2):

* Subjects must have participated in and completed Part 1 per protocol, and have documented assessment attempts for EDSS, T25FW, and 9HPT prior to first open-label dosing.

Key Exclusion Criteria (Part 2):

* Subjects with any significant change in clinical status, including laboratory tests that, in the opinion of the Investigator, would make them unsuitable to participate in this extension study. The Investigator must re-review the subject's medical fitness for participation and consider any diseases that would preclude treatment.
* Subjects who discontinued study treatment in Part 1 OR had fewer than 20 infusions in Part 1 OR missed 2 or more consecutive infusions in Part 1.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 889 (Actual)
Dates: Start 2011-09-13 (Actual); Primary Completion 2015-07-28 (Actual); Study Completion 2016-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (142):
- United States (32):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Lake Barrington, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Burlington, Massachusetts
  - Research Site, Omaha, Nebraska
  - Research Site, Lebanon, New Hampshire
  - Research Site, Teaneck, New Jersey
  - Research Site, Latham, New York
  - Research Site, New York, New York
  - Research Site, Advance, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Uniontown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Clackamas, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Nashville, Tennessee
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Green Bay, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Belgium (3):
  - Research Site, La Louvière
  - Research Site, Melsbroek
  - Research Site, Overpelt
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Czechia (4):
  - Research Site, Hradec Králové, Bohemia
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
- Denmark (5):
  - Research Site, Arthus C
  - Research Site, Esbjerg
  - Research Site, Glostrup Municipality
  - Research Site, København Ø
  - Research Site, Odense
- Finland (3):
  - Research Site, Jyväskylä
  - Research Site, Tampere
  - Research Site, Turku
- France (8):
  - Research Site, Nice, Alpes Maritimes
  - Research Site, Marseille, Bouches-du-Rhône
  - Research Site, Nantes, Loire Atlantique
  - Research Site, Nancy, Meurthe et Moselle
  - Research Site, Lille, Nord
  - Research Site, Bron, Rhone
  - Research Site, Salouël, Somme
  - Research Site, Bordeaux
- Germany (10):
  - Research Site, Bad Mergentheim, Baden-Wurttemberg
  - Research Site, Bad Wilbad, Baden-Wurttemberg
  - Research Site, Tübingen, Baden-Wurttemberg
  - Research Site, Munich, Bavaria
  - Research Site, Hennigsdorf, Brandenburg
  - Research Site, Teupitz, Brandenburg
  - Research Site, Kassel, Hesse
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Münster, North Rhine-Westphalia
  - Research Site, Dresden, Saxony
- Research Site, Dublin, Ireland
- Israel (2):
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
- Italy (12):
  - Research Site, Baggiovara, Modena
  - Research Site, Cefalù, Palermo
  - Research Site, Gallarate, Varese
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Naples
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Pavia
  - Research Site, Rome
- Netherlands (6):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Hoorn
  - Research Site, Nieuwegein
  - Research Site, Sittard-Geleen
- Poland (13):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Plewiska
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Warszawa-Miedzylesie
  - Research Site, Wroclaw
- Russia (5):
  - Research Site, Belgorod
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Tyumen
- Spain (7):
  - Research Site, Barcelona
  - Research Site, El Palmar
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Umeå
- United Kingdom (16):
  - Research Site, Irvine, Ayrshire
  - Research Site, Edgbaston, Birmingham
  - Research Site, Exeter, Devon
  - Research Site, Plymouth, Devon
  - Research Site, London, Greater London
  - Research Site, Hammersmith, London
  - Research Site, Edinburgh, Lothian Region
  - Research Site, Salford, Manchester
  - Research Site, Liverpool, Merseyside
  - Research Site, Norwich, Norfolk
  - Research Site, Nottingham, Nottinghamshire
  - Research Site, Morriston, Swansea
  - Research Site, Newcastle, Tyne
  - Research Site, Brighton
  - Research Site, London
  - Research Site, Sheffield

REFERENCES:
- [Derived] Loomis SJ, Sadhu N, Fisher E, Gafson AR, Huang Y, Yang C, Hughes EE, Marshall E, Herman A, John S, Runz H, Jia X, Bhangale T, Bronson PG. Genome-wide study of longitudinal brain imaging measures of multiple sclerosis progression across six clinical trials. Sci Rep. 2023 Aug 31;13(1):14313. doi: 10.1038/s41598-023-41099-0. PMID 37652990
- [Derived] Beynon V, George IC, Elliott C, Arnold DL, Ke J, Chen H, Zhu L, Ke C, Giovannoni G, Scaramozza M, Campbell N, Bradley DP, Franchimont N, Gafson A, Belachew S. Chronic lesion activity and disability progression in secondary progressive multiple sclerosis. BMJ Neurol Open. 2022 Jun 7;4(1):e000240. doi: 10.1136/bmjno-2021-000240. eCollection 2022. PMID 35720980
- [Derived] Koch MW, Mostert J, Zhang Y, Wolinsky JS, Lublin FD, Strijbis E, Cutter G. Association of Age With Contrast-Enhancing Lesions Across the Multiple Sclerosis Disease Spectrum. Neurology. 2021 Sep 28;97(13):e1334-e1342. doi: 10.1212/WNL.0000000000012603. Epub 2021 Aug 10. PMID 34376508
- [Derived] Kapoor R, Ho PR, Campbell N, Chang I, Deykin A, Forrestal F, Lucas N, Yu B, Arnold DL, Freedman MS, Goldman MD, Hartung HP, Havrdova EK, Jeffery D, Miller A, Sellebjerg F, Cadavid D, Mikol D, Steiner D; ASCEND investigators. Effect of natalizumab on disease progression in secondary progressive multiple sclerosis (ASCEND): a phase 3, randomised, double-blind, placebo-controlled trial with an open-label extension. Lancet Neurol. 2018 May;17(5):405-415. doi: 10.1016/S1474-4422(18)30069-3. Epub 2018 Mar 12. PMID 29545067
- See also: Find out what to expect with TYSABRI MS treatment — http://www.tysabri.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Part 1: participants were randomized to receive placebo intravenously (IV) every 4 weeks for 96 weeks. Part 2: participants transitioned to receive open-label natalizumab 300 mg IV every 4 weeks for at least 96 weeks.
- Natalizumab 300 mg: Part 1: participants were randomized to receive 300 mg of natalizumab IV every 4 weeks for 96 weeks. Part 2: participants transitioned to receive open-label natalizumab 300 mg IV every 4 weeks for at least 96 weeks.
Period: Part 1
Arm/Group | Placebo | Natalizumab 300 mg
Started | 449 | 440
Withdrew Prior to Dosing | 0 | 1
Completed | 312 (Completed Study through Week 108) | 326 (Completed Study through Week 108)
Not Completed | 137 | 114
Not completed — Other | 10 | 24
Not completed — Death | 0 | 1
Not completed — Investigator Decision | 7 | 6
Not completed — Withdrawal by Subject | 74 | 48
Not completed — Lack of Efficacy | 16 | 8
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 15 | 18
Not completed — Ongoing in Follow-Up | 14 | 8
Period: Part 2
Arm/Group | Placebo | Natalizumab 300 mg
Started | 274 | 292
Completed Treatment for 48 Weeks | 98 (completed study treatment for 48 weeks in Part 2) | 111 (completed study treatment for 48 weeks in Part 2)
Completed Treatment for 96 Weeks | 1 (completed study treatment for 96 weeks in Part 2) | 0 (completed study treatment for 96 weeks in Part 2)
Completed Treatment for > 96 Weeks | 1 | 0
Completed | 3 | 6
Not Completed | 271 | 286
Not completed — Adverse Event | 11 | 4
Not completed — Other | 234 | 267
Not completed — Investigator Decision | 6 | 7
Not completed — Withdrawal by Subject | 14 | 5
Not completed — Lack of Efficacy | 4 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who were randomized and received at least 1 infusion of study treatment in Part 1.
Groups:
- Placebo: Part 1: participants were randomized to receive placebo IV every 4 weeks for 96 weeks. Part 2: participants transitioned to receive open-label natalizumab 300 mg IV every 4 weeks for at least 96 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Natalizumab 300 mg | Total
Number analyzed (Participants) | 449 | 439 | 888
Age, Customized [Number; unit: participants]
  20 - 29 years | 10 | 10 | 20
  30 - 39 years | 73 | 50 | 123
  40 - 49 years | 162 | 194 | 356
  ≥ 50 years | 204 | 185 | 389
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 270 | 550
  Male | 169 | 169 | 338

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Confirmed Progression of Disability in One or More of the Expanded Disability Status Scale (EDSS), Timed 25-Foot Walk (T25FW), or 9-Hole Peg Test (9HPT)
Description: Confirmed disability progression, defined as ≥1 of the following criteria (confirmed at a second visit ≥6 months later and at Week 96):
  * Confirmed progression in EDSS (EDSS score increased from baseline [BL] by ≥1 point if BL EDSS ≤5.5 or by ≥0.5 points if BL EDSS ≥6);
  * Confirmed progression in T25FW (T25FW increased by ≥20% of the BL walk);
  * Confirmed progression in 9HPT (9HPT increased by ≥20% of the time taken at BL on either hand and confirmed on the same hand).
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. The T25FW is a quantitative mobility and leg function performance test where the participant is timed while walking for 25 feet. The 9HPT is a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs. The 95% confidence interval (CI) of the percentage is based on normal approximation.
Time Frame: Up to 96 weeks (2 years)
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 448 | 439
percentage of participants
  Confirmed on ≥1 of EDSS, T25FW, or 9HPT at 2 years | 48 [43.1 to 52.4] | 44 [39.8 to 49.1]
  Confirmed on EDSS at 2 years | 15 [11.7 to 18.3] | 16 [12.3 to 19.1]
  Confirmed on T25FW at 2 years | 35 [30.8 to 39.7] | 35 [30.4 to 39.3]
  Confirmed on 9HPT (either hand) at 2 years | 23 [19.3 to 27.1] | 15 [11.3 to 17.9]
  Confirmed on 9HPT (dominant hand) at 2 years | 13 [10.2 to 16.5] | 10 [7.2 to 12.8]
  Confirmed on 9HPT (non-dominant hand) at 2 years | 16 [12.5 to 19.2] | 10 [7.2 to 12.8]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on ≥ 1 of EDSS, T25FW, or 9HPT at 2 years; Test type: Superiority or Other; p = 0.2866, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.66 to 1.13] — active/placebo
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on EDSS; Test type: Superiority or Other; p = 0.7530, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.74 to 1.53] — active/placebo
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on T25FW; Test type: Superiority or Other; p = 0.9137, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.74 to 1.30] — active/placebo
Statistical Analysis 4: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on 9HPT (either hand); Test type: Superiority or Other; p = 0.0012, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.40 to 0.80]
Statistical Analysis 5: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on 9HPT (dominant hand); Test type: Superiority or Other; p = 0.1251, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.48 to 1.09]
Statistical Analysis 6: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on 9HPT (non-dominant hand); Test type: Superiority or Other; p = 0.0091, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.39 to 0.87]

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence that did not necessarily have a causal relationship with this treatment. SAE: any untoward medical occurrence that at any dose: resulted in death; in the view of the Investigator, placed the participant at immediate risk of death (a life-threatening event); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in a congenital anomaly/birth defect. An SAE may have also been any other medically important event in the opinion of the Investigator.
Time Frame: 218 weeks
Population: Safety population: all participants who were randomized in Part 1 and received at least 1 infusion of study treatment in Part 2.
Measure: Number; unit: participants
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 274 | 291
participants
  Any event | 250 | 245
  Moderate or severe event | 157 | 158
  Severe event | 28 | 27
  Related event | 63 | 56
  Serious event | 24 | 39
  Discontinuation of treatment due to event | 12 | 5
  Withdrawal from study due to an event | 11 | 3

3. Secondary Outcome: Part 1: Percentage of Participants With a T25FW Response
Description: T25FW response is defined as any improvement from the best pre-dose T25FW in at least 75% of the scheduled on-treatment visits through Week 96. The T25FW is a quantitative mobility and leg function performance test based on a timed walk over 25 feet. The participant is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. The score for the T25FW is the average of the 2 completed trials. The 95% CI of the percentage is based on normal approximation.
Time Frame: Up to 96 weeks
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment. Excludes participants who withdrew prior to 1 year (defined as stopping treatment prior to Week 48) of participation in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 363 | 383
percentage of participants | 17 [12.7 to 20.3] | 19 [14.6 to 22.4]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Test type: Superiority or Other; p = 0.4369, Regression, Logistic; Based on logistic regression, adjusted for baseline EDSS (<=5.5 or >=6) and T25FW; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.80 to 1.70] — active/placebo

4. Secondary Outcome: Part 1: Change From Baseline in the 12-Item MS Walking Scale (MSWS-12)
Description: MSWS-12 is a participant self-assessment of the walking limitations due to MS during the past 2 weeks. It contains 12 items that measure the impact of MS on walking. Items are summed to generate a total score and transformed to a scale with a range of 0 to 100, where higher scores indicate greater impact on walking. A negative number on change from BL value indicates an improvement in MSWS-12.
Time Frame: Baseline and Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 436 | 431
units on a scale | 4.04 (21.061) | 2.70 (22.110)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Test type: Superiority or Other; p = 0.5409, ANCOVA; p-value for comparison between the active and placebo groups at Week 96 is based on ANCOVA model, adjusted for BL EDSS (<=5.5 or >=6) and BL MSWS-12

5. Secondary Outcome: Part 1: Change From Baseline in Manual Ability Score Based on the ABILHAND Questionnaire
Description: The ABILHAND Questionnaire measures the participant's perceived difficulty in performing everyday manual activities in the last 3 months. The participant completes a 56-item questionnaire by estimating their own difficulty or ease in performing each of 56 activities. Items are summed to generate a total score and transformed to a scale with a range of 0 to 100, where high scores indicate greater impact on manual ability. A positive number on change from baseline value indicates an improvement in ABILHAND.
Time Frame: Baseline and Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 437 | 431
units on a scale | -3.45 (14.739) | -2.44 (13.023)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Test type: Superiority or Other; p = 0.2586, ANCOVA; p-value for comparison between active and placebo groups at Week 96 is based on ANCOVA model, adjusted for BL EDSS (<=5.5 or >=6) and BL ABILHAND

6. Secondary Outcome: Part 1: Change From Baseline in the Multiple Sclerosis Impact Scale-29 Physical (MSIS-29 Physical) Score
Description: The 29-item MSIS-29 is a participant-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a participant's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health. A negative number on change from baseline value indicates an improvement in MSIS-29.
Time Frame: Baseline and Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 428 | 430
units on a scale | 3.34 (20.947) | 0.61 (19.885)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Test type: Superiority or Other; p = 0.1529, ANCOVA; p-value for comparison between active & placebo groups at Wk 96 based on ANCOVA model, adjusted for BL EDSS (≤5.5 or ≥6) & BL MSIS-29 physical score

7. Secondary Outcome: Part 1: Percentage Change From Week 24 in Whole Brain Volume at Week 96
Description: Whole brain volume as measured by MRI.
Time Frame: Week 24 and Week 96
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment. Includes those participants with an assessment at Weeks 24 and 96.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 265 | 287
percentage change | -0.72 (0.656) | -0.66 (0.596)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Only participants with BL brain volume are included in the p-value calculation; Test type: Superiority or Other; p = 0.2424, ANCOVA — natalizumab participants had a baseline after 6 months of treatment and the placebo-to-natalizumab group had a baseline of initiation of treatment; p-value for comparison between active and placebo groups at Week 96 is based on ANCOVA model, adjusted for BL EDSS (<=5.5 or >=6) and BL brain volume

8. Secondary Outcome: Part 1: Percentage of Participants Defined as Confirmed Progressors on EDSS Functional System Scores
Description: The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist. Participants with confirmed progression of disability in EDSS physical functional system scores will be defined as those who met one of the following criteria:
  * an increase of ≥ 1 point from baseline system score of ≥ 1 or an increase of ≥ 2 points from baseline system score of 0 in at least 2 physical functional systems, or
  * an increase of ≥ 2 points from baseline system score of ≥ 1 or an increase of ≥ 3 points from baseline system score of 0 in any 1 physical functional system.
  A confirmed progressor was defined as a participant who met the criteria for disability progression at any given visit and at the 6-Month Confirmation Visit. The 95% CIs are based on normal approximation.
Time Frame: Up to 96 weeks
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 448 | 439
percentage of participants | 29 [25.2 to 33.7] | 25 [20.6 to 28.6]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Test type: Superiority or Other; p = 0.1052, Regression, Logistic; Based on logistic regression, adjusted for baseline EDSS (<=5.5 or >=6); Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.58 to 1.05]

9. Secondary Outcome: Part 2: Percentage of Participants With Disability Worsening at 156 Weeks
Description: Percentage of participants with disability worsening at each scheduled efficacy visit in Part 2, defined as one or more of the following: • ≥ 20% worsening from Part 1 baseline in T25FW; • ≥ 20% worsening from Part 1 baseline in 9HPT; • Worsening from Part 1 baseline in EDSS (≥ 1 point increase if Part 1 baseline EDSS ≤ 5.5 or ≥ 0.5 point increase if Part 1 baseline EDSS > 5.5). The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. The T25FW is a quantitative mobility and leg function performance test where the participant is timed while walking for 25 feet. The 9HPT is a quantitative test of upper extremity function that measures the time it takes to place 9 pegs into 9 holes and then remove the pegs. 95% CIs of percentages are based on normal approximation.
Time Frame: Week 156
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment (Part 2).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 274 | 291
percentage of participants
  Confirmed on ≥1 of EDSS, T25FW, 9HPT at 156 weeks | 61 [55.2 to 66.7] | 52 [45.8 to 57.3]
  Confirmed on EDSS at 156 weeks | 23 [18.3 to 28.4] | 18 [13.8 to 22.6]
  Confirmed on T25FW at 156 weeks | 46 [40.1 to 51.9] | 41 [35.2 to 46.5]
  Confirmed on 9HPT (either hand) at 156 weeks | 28 [23.1 to 33.8] | 19 [14.4 to 23.4]
  Confirmed on 9HPT (dominant hand) at 156 weeks | 18 [13.0 to 22.0] | 12 [8.0 to 15.4]
  Confirmed on 9HPT (non-dominant hand) at 156 weeks | 18 [13.0 to 22.0] | 13 [9.2 to 16.9]
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on ≥ 1 of EDSS, T25FW, or 9HPT at 156 weeks; Test type: Superiority or Other; p = 0.0205, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.47 to 0.94] — active/placebo
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on EDSS at 156 weeks; Test type: Superiority or Other; p = 0.1305, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.48 to 1.10] — active/placebo
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on T25FW at 156 weeks; Test type: Superiority or Other; p = 0.1988, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.57 to 1.12] — active/placebo
Statistical Analysis 4: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on 9HPT (either hand) at 156 weeks; Test type: Superiority or Other; p = 0.0093, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.39 to 0.88] — active/placebo
Statistical Analysis 5: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors onm 9HPT (dominant hand) at 156 weeks; Test type: Superiority or Other; p = 0.0540, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.39 to 1.01] — active/placebo
Statistical Analysis 6: Comparison: Placebo vs Natalizumab 300 mg; Confirmed progressors on 9HPT (non-dominant hand) at 156 weeks; Test type: Superiority or Other; p = 0.1410, Regression, Logistic; Based on logistic regression, adjusted for Baseline EDSS (<=5.5 or >=6) and/or T25FW and/or 9HPT (either hand); Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.44 to 1.12] — active/placebo

10. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 1) in T25FW
Description: The T25FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk. The participant is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. The task is immediately repeated; the score for the T25FW is the average of the two completed trials. Lower scores on time taken to reach 25 foot mark reflect a better outcome. Values are presented for the overall group, as well as the Confirmed Progressor (CP, defined in the primary outcome measure description above) and Non-Progressor (NP) subgroups.
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment (Part 2); n=participants who had an assessment at Baseline and given time point.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 255 | 264
seconds
  Overall: Change from BL to Week 156; n=255, 264 | 12.80 (35.111) | 7.78 (21.251)
  Overall: Change from BL to Week 204; n=39, 38 | 25.01 (56.582) | 9.01 (22.507)
  CP Group: Change from BL to Week 156; n=156, 135 | 21.67 (42.510) | 16.26 (26.943)
  CP Group: Change from BL to Week 204; n=25, 18 | 40.06 (66.275) | 20.89 (28.200)
  NP Group: Change from BL to Week 156; n=99, 129 | -1.17 (3.804) | -1.09 (3.593)
  NP Group: Change from BL to Week 204; n=14, 20 | -1.88 (5.917) | -1.67 (4.613)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Week 156; Test type: Superiority or Other; p = 0.0273, ANCOVA; p-value for comparison between active and placebo at Week 156 based on ANCOVA model, adjusted for BL EDSS (<=5.5 or>=6) and BL T25FW
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.1974, ANCOVA; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.2506, ANCOVA; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in T25FW
Description: The T25FW is a quantitative mobility and leg function performance test based on a timed 25-foot walk. The participant is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the participant has reached the 25-foot mark. The task is immediately repeated; the score for the T25FW is the average of the two completed trials. Values are presented for the overall group, as well as the CP (defined in the primary outcome measure description above) and NP subgroups.
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 255 | 264
percentage change
  Overall: Change from BL at Week 156; n=255, 264 | 75.52 (166.191) | 55.91 (130.286)
  Overall: Change from BL at Week 204; n=39, 38 | 130.72 (272.117) | 71.09 (177.668)
  CP Group: Change from BL at Week 156; n=156, 135 | 127.05 (195.138) | 113.51 (160.857)
  CP Group: Change from BL at Week 204; n=25, 18 | 206.78 (316.344) | 158.91 (228.458)
  NP Group: Change from BL at Week 156; n=99, 129 | -5.68 (21.708) | -4.37 (25.050)
  NP Group: Change from BL at Week 204; n=14, 20 | -5.09 (26.591) | -7.94 (29.856)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Overall: Week 156; Test type: Superiority or Other; p = 0.0960, ANCOVA; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.4957, ANCOVA; [statistical method as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.2916, ANCOVA; [statistical method as in outcome 10, analysis 1]

12. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 1) in 9HPT (Dominant Hand)
Description: The 9HPT is a brief, standardized, quantitative test of upper extremity function. The participant picks up 9 pegs puts them in a block containing nine empty holes, and, once they are in the holes, removes them again as quickly as possible one at a time. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The two trials for each hand are averaged. Values are presented for the overall group, as well as the CP (defined in the primary outcome measure description above) and NP subgroups.
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 257 | 271
seconds
  Overall: Change from BL to Week 156; n= 257, 271 | 5.22 (27.728) | 2.12 (16.719)
  Overall: Change from BL to Week 204; n=39, 38 | 0.56 (7.923) | 2.65 (16.001)
  CP Group: Change from BL to Week 156; n=158, 138 | 10.12 (33.675) | 5.01 (20.625)
  CP Group: Change from BL to Week 204; n=24, 19 | 2.36 (9.187) | 6.03 (21.994)
  NP Group: Change from BL to Week 156; n=99, 133 | -2.60 (9.543) | -0.89 (10.602)
  NP Group: Change from BL to Week 204; n=15, 19 | -2.32 (4.153) | -0.73 (4.292)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Overall, Week 156; Test type: Superiority or Other; p = 0.1119, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA model, adjusted for BL EDSS (≤5.5 or ≥6) & BL 9HPT (dominant hand)
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.1129, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.2351, ANCOVA; [statistical method as in outcome 12, analysis 1]

13. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in 9HPT (Dominant Hand)
Description: as for outcome 12
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 257 | 271
percentage change
  Overall: Change from BL to Week 156; n=257, 271 | 14.32 (59.727) | 5.25 (32.649)
  Overall: Change from BL to Week 204; n=39, 38 | 2.27 (19.193) | 6.87 (32.333)
  CP Group: Change from BL to Week 156; n=158, 138 | 25.87 (72.621) | 12.84 (40.232)
  CP Group: Change from BL to Week 204; n=24, 19 | 8.43 (20.247) | 16.25 (41.317)
  NP Group: Change from BL to Week 156; n=99, 133 | -4.10 (17.661) | -2.63 (19.436)
  NP Group: Change from BL to Week 204; n=15, 19 | -7.57 (12.560) | -2.52 (15.998)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Overall: Week 156; Test type: Superiority or Other; p = 0.0261, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.0585, ANCOVA; [statistical method as in outcome 12, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.6095, ANCOVA; [statistical method as in outcome 12, analysis 1]

14. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 1) in 9HPT (Non-Dominant Hand)
Description: as for outcome 12
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 254 | 269
seconds
  Overall: Change from BL to Week 156; n=254, 269 | 5.24 (32.910) | 4.62 (30.333)
  Overall: Change from BL to Week 204; n=40, 40 | 1.41 (16.952) | 4.91 (33.808)
  CP Group: Change from BL to Week 156; n=155, 137 | 11.25 (39.513) | 11.25 (38.296)
  CP Group: Change from BL to Week 204; n=25, 20 | 5.87 (17.474) | 17.20 (34.632)
  NP Group: Change from BL to Week 156; n=99, 132 | -4.17 (13.999) | -2.26 (16.311)
  NP Group: Change from BL to Week 204; n=15, 20 | -6.04 (13.491) | -7.39 (28.780)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Overall: Week 156; Test type: Superiority or Other; p = 0.7230, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA, adjusted for BL EDSS (≤5.5 or ≥6) & BL 9HPT (non-dominant hand)
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.8781, ANCOVA; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.2751, ANCOVA; [statistical method as in outcome 14, analysis 1]

15. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in 9HPT (Non-Dominant Hand)
Description: as for outcome 12
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 254 | 269
percentage change
  Overall: Change from BL to Week 156; n=254, 269 | 13.87 (64.959) | 11.04 (47.942)
  Overall: Change from BL to Week 204; n=40, 40 | 3.67 (28.755) | 18.57 (62.537)
  CP Group: Change from BL to Week 156; n=155, 137 | 26.33 (79.957) | 23.51 (60.074)
  CP Group: Change from BL to Week 204; n=25, 20 | 11.87 (31.050) | 43.12 (80.639)
  NP Group: Change from BL to Week 156; n=99, 132 | -5.63 (14.765) | -1.89 (24.987)
  NP Group: Change from BL to Week 204; n=15, 20 | -9.98 (18.188) | -5.98 (16.005)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Overall: Week 156; Test type: Superiority or Other; p = 0.5051, ANCOVA; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.7283, ANCOVA; [statistical method as in outcome 14, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.1666, ANCOVA; [statistical method as in outcome 14, analysis 1]

16. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 1) in EDSS
Description: The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist. Values are presented for the overall group, as well as the CP (defined in the primary outcome measure description above) and NP subgroups.
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 260 | 275
units on a scale
  Overall: Change from BL to Week 156; n=260, 275 | 0.11 (0.746) | 0.06 (0.797)
  Overall: Change from BL to Week 204; n=40, 40 | -0.01 (0.895) | 0.15 (0.928)
  CP Group: Change from BL to Week 156; n=162, 141 | 0.38 (0.631) | 0.36 (0.703)
  CP Group: Change from BL to Week 204; n=25, 20 | 0.28 (0.542) | 0.68 (0.634)
  NP Group: Change from BL to Week 156; n=98, 134 | -0.33 (0.718) | -0.25 (0.775)
  NP Group: Change from BL to Week 204; n=15, 20 | -0.50 (1.150) | -0.38 (0.887)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Overall: Week 156; Test type: Superiority or Other; p = 0.4330, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA, adjusted for BL EDSS (≤5.5 or ≥6)
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.7122, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA, adjusted for BL EDSS (≤5.5 or ≥6)
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.3861, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA, adjusted for BL EDSS (≤5.5 or ≥6)

17. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in EDSS
Description: as for outcome 16
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 260 | 275
percentage change
  Overall: Change from BL to Week 156; n=260, 275 | 2.07 (15.188) | 1.65 (16.530)
  Overall: Change from BL to Week 204; n=40, 40 | -0.63 (17.889) | 2.91 (18.656)
  CP Group Change from BL to Week 156; n=162, 141 | 7.23 (13.513) | 7.30 (15.728)
  CP Group Change from BL to Week 204; n=25, 20 | 5.31 (10.711) | 13.18 (13.957)
  NP Group Change from BL to Week 156; n=98, 134 | -6.47 (13.951) | -4.29 (15.266)
  NP Group Change from BL to Week 204; n=15, 20 | -10.53 (22.953) | -7.35 (17.260)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Overall: Week 156; Test type: Superiority or Other; p = 0.7225, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA, adjusted for BL EDSS (≤5.5 or ≥6)
Statistical Analysis 2: Comparison: Placebo vs Natalizumab 300 mg; CP Group: Week 156; Test type: Superiority or Other; p = 0.9121, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA, adjusted for BL EDSS (≤5.5 or ≥6)
Statistical Analysis 3: Comparison: Placebo vs Natalizumab 300 mg; NP Group: Week 156; Test type: Superiority or Other; p = 0.2594, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA, adjusted for BL EDSS (≤5.5 or ≥6)

18. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 1) in the 6-Minute Walk Test (6MWT)
Description: The 6MWT measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Frame: Baseline (Part 1) and Weeks 156 and 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 272 | 290
meters
  Change from BL to Week 156; n=272, 289 | -32.1 (117.55) | -40.4 (219.60)
  Change from BL to Week 204; n=272, 290 | -33.3 (119.40) | -40.7 (219.58)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Week 156; Test type: Superiority or Other; p = 0.8066, ANCOVA; p-value for comparison between active & placebo groups at Week 156 based on ANCOVA model, adjusted for BL EDSS (≤5.5 or ≥6) & BL 6MWT

19. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in the 6MWT
Description: as for outcome 18
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: Actual change from baseline tables are provided in previous Outcome Measure. Due to the nature of self-selected population in an extension trial and sparse data on Weeks 204 and 252, further tabulations on percentage changes on these endpoints were deemed less meaningful and unnecessary.
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 1) in the MSIS-29 Physical Score
Description: The 29-item MSIS-29 is a patient-reported outcome measure to assess the impact of MS on day-to-day life during the past 2 weeks from a patient's perspective; it measures 20 physical items and 9 psychological items. The physical score is generated by summing individual items and then transforming to a scale with a range of 0 to 100, where high scores indicate worse health. A negative number on change from baseline value indicates an improvement in MSIS-29.
Time Frame: Baseline (Part 1) and Weeks 156 and 204
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment (Part 2) who had an assessment at Baseline and given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 274 | 291
units on a scale
  Change from BL to Week 156 | 0.32 (20.943) | 0.05 (20.843)
  Change to from BL Week 204 | 0.91 (21.018) | -0.28 (20.596)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Test type: Superiority or Other; p = 0.7084, ANCOVA; p-value for comparison between active & placebo at Week 156 based on ANCOVA model, adjusted for BL EDSS (≤5.5 or ≥6) & BL MSIS-29 physical score

21. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in the MSIS-29 Physical Score
Description: as for outcome 20
Time Frame: Baseline (Part 1) and Weeks 156, 204
Population: as for outcome 19
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 1) in the Symbol Digit Modalities Test (SDMT)
Description: SDMT is a screening test for cognitive impairment. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 to 110 (best).
Time Frame: Baseline (Part 1) and every 4 weeks from Week 108 to Week 204
Population: Intent to treat population: all participants who were randomized and received at least 1 infusion of study treatment (Part 2). Missing values were imputed using last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 273 | 291
units on a scale
  Change from BL to Week 108 | 13.6 (14.19) | 15.5 (13.82)
  Change from BL to Week 112 | 14.4 (13.72) | 15.1 (13.50)
  Change from BL to Week 116 | 14.1 (13.84) | 15.3 (13.51)
  Change from BL to Week 120 | 14.3 (14.23) | 15.3 (13.68)
  Change from BL to Week 124 | 14.4 (14.02) | 15.7 (13.69)
  Change from BL to Week 128 | 15.1 (14.49) | 15.7 (13.72)
  Change from BL to Week 132 | 15.1 (14.52) | 15.6 (13.63)
  Change from BL to Week 136 | 14.8 (14.56) | 16.3 (13.75)
  Change from BL to Week 140 | 15.4 (14.98) | 16.4 (14.29)
  Change from BL to Week 144 | 15.7 (15.23) | 16.2 (14.22)
  Change from BL to Week 148 | 15.5 (15.34) | 16.3 (14.35)
  Change from BL to Week 152 | 15.5 (14.98) | 16.3 (14.25)
  Change from BL to Week 156 | 11.2 (13.10) | 12.3 (14.59)
  Change from BL to Week 160 | 15.2 (14.92) | 16.2 (14.61)
  Change from BL to Week 164 | 15.6 (15.21) | 16.3 (14.64)
  Change from BL to Week 168 | 15.8 (15.52) | 16.4 (14.78)
  Change from BL to Week 172 | 15.6 (15.40) | 16.3 (14.64)
  Change from BL to Week 176 | 15.5 (15.58) | 16.3 (14.91)
  Change from BL to Week 180 | 15.5 (15.23) | 16.4 (14.89)
  Change from BL to Week 184 | 15.6 (15.34) | 16.3 (14.81)
  Change from BL to Week 188 | 15.6 (15.38) | 16.4 (14.77)
  Change from BL to Week 192 | 15.6 (15.46) | 16.3 (14.79)
  Change from BL to Week 196 | 15.7 (15.45) | 16.3 (14.69)
  Change from BL to Week 200 | 15.7 (15.47) | 16.3 (14.69)
  Change from BL to Week 204 | 15.7 (15.43) | 16.3 (14.69)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Week 156; Test type: Superiority or Other; p = 0.3465, ANCOVA; p-value for comparison between active and placebo at Week 156 based on ANCOVA model, adjusted for BL EDSS (<=5.5 or>=6) and BL SDMT

23. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in the SDMT
Description: as for outcome 22
Time Frame: Baseline (Part 1) and every 4 weeks from Week 108 to Week 204
Population: Actual change from baseline tables are provided in previous Outcome Measure. Due to the nature of self-selected population in an extension trial and sparse data up to Weeks 204 and 252, further tabulations on percentage changes on these endpoints were deemed less meaningful and unnecessary, and the analysis was not done.
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Part 2: Absolute Change From Baseline (Part 2) in the Work Productivity and Activity Impairment - Multiple Sclerosis (WPAI-MS) Questionnaire
Description: The WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (percentage of work time missed) 2. Presenteesism (percentage of impairment at work/reduced on-the-job effectiveness) 3. Work productivity loss (percentage of overall work impairment [absenteeism plus presenteeism]) 4. Activity Impairment (percentage of overall activity impairment). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Part 2 Baseline (Week 108) and Weeks 156 and 204
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 272 | 291
percentage of impairment
  Absenteeism: Week 108 | 2.6 (12.80) | 1.4 (8.24)
  Absenteeism: Week 156 | 3.0 (14.61) | 4.1 (17.36)
  Absenteeism: Week 204 | 3.0 (14.61) | 4.2 (16.89)
  Presenteeism: Week 108 | 30.6 (12.10) | 30.9 (11.71)
  Presenteeism: Week 156 | 30.8 (12.17) | 33.0 (14.23)
  Presenteeism: Week 204 | 31.0 (12.29) | 32.2 (13.78)
  Work Productivity Loss: Week 108 | 30.9 (12.36) | 31.2 (11.70)
  Work Productivity Loss: Week 156 | 31.6 (13.54) | 33.9 (15.75)
  Work Productivity Loss: Week 204 | 31.9 (13.66) | 33.3 (15.61)
  Activity Impairment: Week 108 | 56.1 (24.78) | 58.0 (24.84)
  Activity Impairment: Week 156 | 56.8 (26.49) | 58.5 (24.08)
  Activity Impairment: Week 204 | 57.2 (25.15) | 59.8 (23.60)

25. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 2) in the WPAI-MS Questionnaire
Description: The WPAI questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (percentage of work time missed) 2. Presenteesism (percentage of impairment at work/reduced on-the-job effectiveness) 3. Work productivity loss (WPL; percentage of overall work impairment [absenteeism plus presenteeism]) 4. Activity Impairment (AI; percentage of overall activity impairment). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Time Frame: Part 2 Baseline (Week 108) and Weeks 156 and 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 274 | 291
percentage change
  Absenteeism: Change at Week 156; n=18,17 | -10.3 (116.81) | -7.4 (95.77)
  Absenteeism: Change at Week 204; n=18, 17 | -6.6 (116.90) | 151.5 (457.29)
  Presenteeism: Change at Week 156; n=264, 285 | 4.0 (50.08) | 14.4 (90.39)
  Presenteeism: Change at Week 204; n=264, 285 | 5.3 (51.23) | 7.4 (58.95)
  WPL: Change at Week 156; n=264,286 | 4.7 (51.73) | 16.8 (95.43)
  WPL: Change at Week 204; n=264, 286 | 5.9 (53.44) | 10.6 (69.34)
  AI: Change at Week 156; n=264, 284 | 16.0 (95.68) | 15.7 (83.70)
  AI: Change at Week 204; n=264, 284 | 16.1 (88.56) | 20.4 (99.54)

26. Secondary Outcome: Part 2: Percentage Change From Week 24 (Part 1) in Whole Brain Volume
Description: Whole brain volume as measured by MRI.
Time Frame: Week 24 (Part 1) and Weeks 156 and 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 274 | 291
percentage change
  Change from Week 24 to Week 156; n=155, 175 | -1.164 (0.8228) | -0.948 (0.7193)
  Change from Week 24 to Week 204; n=28, 24 | -1.687 (1.2872) | -1.517 (0.8412)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Percentage change from Week 24 to Week 156; Test type: Superiority or Other; p = 0.0070, ANCOVA — [p-value comment as in outcome 7, analysis 1]; p-value for comparison between active & placebo at Week 156 based on ANCOVA model, adjusted for BL EDSS (≤5.5 or ≥6) & BL normalized brain volume

27. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in Whole Gray Matter Brain Volume
Description: Whole grey matter brain volume as measured by MRI.
Time Frame: Baseline (Part 1) and Weeks 156 and 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 274 | 291
percentage change
  Change from Baseline to Week 156; n=149, 170 | -1.566 (0.9303) | -1.514 (0.8969)
  Change from Baseline to Week 204; n=26, 20 | -1.883 (1.4222) | -2.086 (0.9068)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Percentage hange from Baseline to Week 156; Test type: Superiority or Other; p = 0.5034, ANCOVA — [p-value comment as in outcome 7, analysis 1]; p-value for comparison between active & placebo at Week 156 based on ANCOVA model, adjusted for BL EDSS (≤5.5 or ≥6) & BL WGM brain volume

28. Secondary Outcome: Part 2: Summary of New/Enlarging T2 Lesion Counts
Description: New or enlarging T2 lesions as measured by MRI.
Time Frame: Baseline (Part 1) up to Week 204
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 274 | 291
lesions
  At Week 24 compared to BL; n=272, 287 | 2.1 (4.24) | 0.6 (3.27)
  At Week 48 compared to Week 24; n=272, 289 | 1.8 (4.47) | 0.0 (0.37)
  At Week 72 compared to Week 48; n=271, 287 | 1.6 (3.76) | 0.0 (0.19)
  At Week 96 compared to Week 72; n=269, 284 | 1.8 (4.33) | 0.0 (0.00)
  At Week 108 compared to Week 96; n=269, 288 | 1.2 (3.38) | 0.0 (0.13)
  At Week 156 compared to Week 108; n=245, 258 | 0.2 (0.79) | 0.0 (0.20)
  At Week 204 compared to Week 156; n=50, 47 | 0.0 (0.20) | 0.0 (0.15)
  Cumulative count from BL to Week 204; n=274, 291 | 8.6 (16.04) | 0.7 (3.53)
Statistical Analysis 1: Comparison: Placebo vs Natalizumab 300 mg; Week 156; Test type: Superiority or Other; p < 0.0001, negative binomial regression model — p-value for comparison between the active and placebo groups at Week 156 compared to Week 108 is based on negative binomial regression model, adjusted for baseline EDSS (<=5.5 or >=6) and baseline volume of T2 lesions; natalizumab participants had a baseline after 6 months of treatment and the placebo-to-natalizumab group had a baseline of initiation of treatment

29. Secondary Outcome: Part 2: Percentage Change From Baseline (Part 1) in Number of New/Enlarging T2 Lesions
Description: New or enlarging T2 lesions as measured by MRI.
Time Frame: Baseline (Part 1) and Weeks 156 and 204
Population: Summary new/enlarging T2 lesion values are provided in previous Outcome Measure. Due to the nature of self-selected population in an extension trial and sparse data up to Week 204, further tabulations on percentage changes on these endpoints were deemed less meaningful and unnecessary, and the analysis was not done.
Arm/Group | Placebo | Natalizumab 300 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are captured through the last study visit; participants were followed through Week 228, or 24 weeks following last dose of study treatment, or premature withdrawal.
Description: Treatment-emergent adverse events only are presented.
Arm/Group | Placebo | Natalizumab 300 mg
Serious Adverse Events (participants affected / at risk) | 100/449 | 90/439
Other Adverse Events (participants affected / at risk) | 347/449 | 325/439
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=449) | Natalizumab 300 mg (N=439)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Pelvic kidney (Congenital, familial and genetic disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 2
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 3
Anaphylactic shock (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 2 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 3
H1n1 influenza (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 5 | 2
Prostatic abscess (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 12 | 5
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Ear injury (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral venous thrombosis (Nervous system disorders) | 0 | 1
Cervical myelopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 5 | 0
Multiple sclerosis relapse (Nervous system disorders) | 28 | 21
Muscle spasticity (Nervous system disorders) | 0 | 2
Optic neuritis (Nervous system disorders) | 2 | 0
Quadriparesis (Nervous system disorders) | 1 | 0
Secondary progressive multiple sclerosis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tonic convulsion (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Uhthoff's phenomenon (Nervous system disorders) | 3 | 1
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Joint surgery (Surgical and medical procedures) | 0 | 1
Limb operation (Surgical and medical procedures) | 0 | 1
Meniscus operation (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=449) | Natalizumab 300 mg (N=439)
Constipation (Gastrointestinal disorders) | 26 | 21
Diarrhoea (Gastrointestinal disorders) | 31 | 33
Nausea (Gastrointestinal disorders) | 23 | 34
Fatigue (General disorders) | 53 | 59
Cystitis (Infections and infestations) | 16 | 22
Influenza (Infections and infestations) | 33 | 32
Nasopharyngitis (Infections and infestations) | 73 | 98
Upper respiratory tract infection (Infections and infestations) | 30 | 48
Urinary tract infection (Infections and infestations) | 103 | 100
Contusion (Injury, poisoning and procedural complications) | 17 | 26
Fall (Injury, poisoning and procedural complications) | 85 | 82
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 43
Back pain (Musculoskeletal and connective tissue disorders) | 50 | 45
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 23
Muscular weakness (Musculoskeletal and connective tissue disorders) | 39 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 42 | 42
Dizziness (Nervous system disorders) | 35 | 22
Headache (Nervous system disorders) | 50 | 66
Multiple sclerosis relapse (Nervous system disorders) | 116 | 68
Muscle spasticity (Nervous system disorders) | 27 | 17
Paraesthesia (Nervous system disorders) | 13 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.